CLINICAL TRIAL: NCT02560649
Title: A Prospective, Randomized, Multicenter, Open-label, Exploratory Study of Utilizing of "Response-Guided-Therapy (RGT)" Strategy on Optimal Nucleoside Analogue (NUC)-Experienced Patients
Brief Title: An Exploratory Study of RGT Strategy on Optimal NUC-experienced Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Qing XIe, director of infectious disease, Ruijin Hospital
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: PYRAMID
Record Dates: First submitted 2015-09-22; First posted 2015-09-25 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a; entecavir; Lamivudine; lipoarabinomannan; adefovir; Tenofovir

ARMS (3):
- A:PEG+NUC (HBsAg<200IU/ml at week 24) (Experimental): Peginterferon alfa-2a 180μg /wk plus nucleoside analogue(NUC):
  HBsAg<200IU/ml at week 24 (Following treatment with Peginterferon alfa-2a plus nucleoside analogue(NUC) for 24 weeks)
  Interventions: Drug: Peginterferon alfa-2a plus Entecavir; Drug: Peginterferon alfa-2a plus Lamivudine; Drug: Peginterferon alfa-2a plus Adefovir; Drug: Peginterferon alfa-2a plus Tenofovir
- B:PEG+NUC(HBsAg>200IU/ml at week 24) (Active Comparator): Peginterferon alfa-2a 180μg /wk plus+nucleoside analogue(NUC):
  HBsAg>200IU/ml at week 24 (Following treatment with Peginterferon alfa-2a plus nucleoside analogue(NUC) for 24 weeks)
  Interventions: Drug: Peginterferon alfa-2a plus Entecavir; Drug: Peginterferon alfa-2a plus Lamivudine; Drug: Peginterferon alfa-2a plus Adefovir; Drug: Peginterferon alfa-2a plus Tenofovir
- C:NUC(HBsAg>200IU/ml at week 24) (Active Comparator): nucleoside analogue(NUC):
  HBsAg>200IU/ml at week 24 (Following treatment with Peginterferon alfa-2a plus nucleoside analogue(NUC) for 24 weeks)
  Interventions: Drug: Entecavir; Drug: Lamivudine; Drug: Adefovir; Drug: Tenofovir disoproxil

INTERVENTIONS:
Drug: Peginterferon alfa-2a plus Entecavir — Peginterferon alfa-2a 180μg /wk plus Entecavir 0.5mg qd for 48 weeks(Arm A and B)
  Other Names: Pegasys; ETV
  Arms: A:PEG+NUC (HBsAg<200IU/ml at week 24); B:PEG+NUC(HBsAg>200IU/ml at week 24)
Drug: Peginterferon alfa-2a plus Lamivudine — Peginterferon alfa-2a 180μg /wk plus Lamivudine 0.1g qd for 48 weeks(Arm A and B)
  Other Names: Pegasys; LAM
  Arms: A:PEG+NUC (HBsAg<200IU/ml at week 24); B:PEG+NUC(HBsAg>200IU/ml at week 24)
Drug: Peginterferon alfa-2a plus Adefovir — Peginterferon alfa-2a 180μg /wk plus Adefovir 10mg qd for 48 weeks(Arm A and B)
  Other Names: Pegasys;ADV
  Arms: A:PEG+NUC (HBsAg<200IU/ml at week 24); B:PEG+NUC(HBsAg>200IU/ml at week 24)
Drug: Peginterferon alfa-2a plus Tenofovir — Peginterferon alfa-2a 180μg /wk plus Tenofovir 300mg qd for 48 weeks(Arm A and B)
  Other Names: Pegasys;TDF
  Arms: A:PEG+NUC (HBsAg<200IU/ml at week 24); B:PEG+NUC(HBsAg>200IU/ml at week 24)
Drug: Entecavir — Entecavir 0.5mg qd for 24 weeks(Arm C)
  Other Names: ETV
  Arms: C:NUC(HBsAg>200IU/ml at week 24)
Drug: Lamivudine — Lamivudine 0.1g qd for 24 weeks(Arm C)
  Other Names: LAM
  Arms: C:NUC(HBsAg>200IU/ml at week 24)
Drug: Adefovir — Adefovir 10mg qd for 24 weeks(ArmC)
  Other Names: Adefovir dipivoxil;ADV
  Arms: C:NUC(HBsAg>200IU/ml at week 24)
Drug: Tenofovir disoproxil — Tenofovir 300mg qd for 24 weeks(Arm C)
  Other Names: Tenofovir disoproxil;TDF
  Arms: C:NUC(HBsAg>200IU/ml at week 24)

SUMMARY:
The aim of current study is to investigate whether the HBsAg clearance rate can be improved if applying RGT((Response-Guided Therapy) strategy in HBeAg positive CHB(chronic hepatitis B) patients treated by nucleoside analogue(NUC) achieved HBVDNA<1000copies/ml，and HBsAg<5000IU/ml; &HBeAg<100PEIU/ml (or470s/co), combined with PEG-IFN a-2a for 24 weeks.

DETAILED DESCRIPTION:
The current study is a prospective, randomized, open, multi-center investigation. The aim of current study is to investigate whether the HBsAg clearance rate can be improved if applying RGT strategy in HBeAg positive CHB patients treated by NUC achieved HBVDNA<1000copies/ml，and HBsAg<5000IU/ml; &HBeAg<100PEIU/ml (or470s/co), combined with PEG-IFN a-2a for 24 weeks. Then the subjects will be divided into three groups according to qHBsAg levels of week 24 (RGT). For the subjects who qHBsAg<200IU/ml of week 24, they are defined in Group A; the subjects in Group A will continue to be treated by NUC combined with PEG-IFN a-2a 180μg for another 24 weeks(total will be 48 weeks). If the qHBsAg at week 24 did not achieve minor 200IU/ml, the subjects will be randomized to 2 groups: Group B: the subjects will continue to be treated by NUC combined with PEG-IFN a-2a 180μg for another 24 weeks (total will be 48 weeks); Group C: the subjects will be treated by NUC until 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients with age ≥18 and ≤65 years;
2. There should be evidences that HBsAg and HBeAg have been positive for more than 6 months with HBsAb and HBeAb negative before treated with nucleoside analogue(NUC) (except of telbivudine);
3. Treated with NUC (except of telbivudine)for more than 24 weeks and achieve HBV DNA<1000copies/ml and HBsAg<5000IU/ml；&HBeAg<100PEIU/ml(470s/co);
4. Without contra-indications to Peginterferon alfa-2a therapy as detailed in the label;
5. Without co-infection with hepatitis C, hepatitis D and HIV;
6. Women without ongoing pregnancy or breast feeding and willing to take an effective contraceptive measure during the treatment
7. Agree to participate in the study and sign the patient informed consent form.

Exclusion criteria

1. Co-infection with active hepatitis A, hepatitis C, hepatitis D and/or human immunodeficiency virus (HIV)
2. AFP(alpha fetoprotein)>50ng/ml and/or evidence of hepatocellular carcinoma
3. Evidence of decompensated liver disease (Child-Pugh scores >5). Child-Pugh >5 means that, if one of the following 6 conditions is met, the patient has to be excluded:

   * Serum albumin <35 g/L
   * Prothrombin time prolonged≥ 4 seconds or PTA(prothrombin activity) < 60%
   * Serum bilirubin > 34 µmol/L
   * History of encephalopathy
   * Ascites
4. History or other evidence of a medical condition associated with chronic liver disease other than viral hepatitis (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures, thalassemia)
5. Pregnant or breast-feeding Women
6. ANC(absolute neutrophil count)<1.5x 10^9/L or PLT(platelet count)<90x 10^9/L
7. Consuming alcohol in excess of 20g/day for women and 30g/day for men within 6 months prior to enrollment
8. History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as major depression or psychosis that treated with antidepressant medication or a major tranquilizer at therapeutic doses respectively at any time prior to 3 months or any history of the following: a suicidal attempt hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease
9. History of immunologically mediated disease, (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, rheumatoid arthritis etc.)
10. History of esophageal varices bleeding or other evidence of esophageal varices bleeding or other symptoms consistent with decompensated liver disease
11. History of chronic pulmonary disease associated with functional limitation
12. History of severe cardiac disease (e.g., NYHA Functional Class III or IV, myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina or other significant cardiovascular diseases)
13. Hemodialysis patients or patients with renal insufficiency
14. History of a severe seizure disorder or current anticonvulsant use
15. Major organ transplantation or other evidence of severe illness, malignancy, or any other conditions, which would make the patient, in the opinion of the investigator, unsuitable for the study
16. History of thyroid disease poorly controlled on prescribed medications
17. Evidence of severe retinopathy or clinically relevant ophthalmologic disorder
18. History of other severe disease or evidence of other severe disease or any other illness or conditions that the investigator believe that patients are not suitable to join in the study
19. Immunomodulatory treatment (including interferon) or LDT(telbivudine) within 1 year prior to the first dose of treatment
20. Patients included in another trial or having been given investigational drugs within 12 weeks prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-08 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants who achieve HBsAg clearance | Week 48
  To investigate whether HBsAg clearance rate can be improved at week 48 following applying RGT strategy(week 24) in NUC-experience subjects will be measured by the number of participants who achieve HBsAg clearance

SECONDARY OUTCOMES:
Number of participants who achieve HBsAg seroconversion | Week 48
  To investigate the HBsAg seroconversion rate at week 48 can be improved following applying RGT strategy in NUC-experience subjects will be measured by the number of participants who achieve HBsAg seroconversion
Number of participants who achieve HBeAg loss | Week 48
  To investigate the HBeAg loss rate at week 48 can be improved following applying RGT strategy in NUC-experience subjects will be measured by the number of participants who achieve HBeAg loss
Number of participants who achieve HBeAg seroconversion | Week 48
  To investigate the HBeAg seroconversion rate at week 48 will be improved following applying RGT strategy in NUC-experience subjects will be measured by the number of participants who achieve HBeAg seroconversion
Percentage of of participants who achieve HBsAg decline >2log from baseline(0 week) | Week 48
  To investigate HBsAg decline from baseline at week 48 following applying RGT strategy in NUC-experience subjects by measured the percentage of of participants who achieve HBsAg decline>2log from baseline(0 week)
Percentage of of participants who achieve HBsAg <10IU/mL | Week 48
  To investigate the percentage of of participants who achieve HBsAg <100IU/mLat week 48 following applying RGT strategy in NUC-experience subjects
Percentage of of participants who achieve combined response(defined as HBeAg seroconversion and HBVDNA<300copies/mL) | Week 48
  To investigate the percentage of of participants who achieve combined response at week 48 following applying RGT strategy in NUC-experience subjects will be measured by number of participants who achieve combined response
Percentage of of participants who achieve dural response I (defined as HBeAg seroconversion and HBsAg<100IU/mL) | Week 48
  To investigate the percentage of of participants who achieve dural response I at week 48 following applying RGT strategy in NUC-experience subjects will be measured by number of participants who achieve dural response
Percentage of of participants who achieve dural response II (defined as HBeAg seroconversion and HBsAg<10IU/mL) | Week 48
  To investigate the percentage of of participants who achieve dural response II at week 48 following applying RGT strategy in NUC-experience subjects will be measured by number of participants who achieve dural response
Number of participants who relapses (HBVDNA>1000copies/ml) | Week 48
  To investigate the number of participants who relapses following applying RGT strategy in NUC-experience subjects
Number of Participants with AE | Week 48
  Number of participants with adverse events as a measure of safety and tolerability
Number of Participants with SAE | Week 48
  Number of participants with SAEs as a measure of safety and tolerability

REFERENCES:
- [Background] Ning Q, Han M, Sun Y, Jiang J, Tan D, Hou J, Tang H, Sheng J, Zhao M. Switching from entecavir to PegIFN alfa-2a in patients with HBeAg-positive chronic hepatitis B: a randomised open-label trial (OSST trial). J Hepatol. 2014 Oct;61(4):777-84. doi: 10.1016/j.jhep.2014.05.044. Epub 2014 Jun 7. PMID 24915612
- [Background] P. Hu et al. 2015 EASL abstract O116. PREDICTIVE VALUE OF BASELINE AND ON-TREATMENT qHBsAg LEVEL IN HBeAg POSITIVE CHB PATIENTS WHO SWITCHED FROM NUCS TO PEGYLATED INTERFERON A-2A: A FURTHER ANALYSIS FROM NEW SWITCH STUDY
- [Background] Brouwer WP, Xie Q, Sonneveld MJ, Zhang N, Zhang Q, Tabak F, Streinu-Cercel A, Wang JY, Idilman R, Reesink HW, Diculescu M, Simon K, Voiculescu M, Akdogan M, Mazur W, Reijnders JG, Verhey E, Hansen BE, Janssen HL; ARES Study Group. Adding pegylated interferon to entecavir for hepatitis B e antigen-positive chronic hepatitis B: A multicenter randomized trial (ARES study). Hepatology. 2015 May;61(5):1512-22. doi: 10.1002/hep.27586. Epub 2015 Feb 27. PMID 25348661